CLINICAL TRIAL: NCT05126706
Title: Validating Efficacy for Digital Lifestyle Management for Weight Loss Control After Thyroidectomy in Thyroid Cancer Patients
Brief Title: Digital Lifestyle Management for Weight Loss Control After Thyroidectomy in Thyroid Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kyu Eun Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2105-192-1224
Record Dates: First submitted 2021-09-26; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Weight Change, Body
Keywords: Digital lifestyle management; Thyroid cancer; Total thyroidectomy; Obesity
MeSH Terms: conditions — Body Weight Changes; Thyroid Neoplasms; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital lifestyle management group (Experimental): In the experimental group (digital lifestyle management group), 54 patients are randomly assigned to the digital lifestyle management group. The patients use this application for the first 4 months with Noom applications with 1:1 personalized coaching intervention, and then, use this app by self-help program without coaching intervention. In order to monitor the psychological state of the patients, all the patients are given daily assessment online questionnaires and additional questionnaires to evaluate the quality of life at the baseline, 4 months, and 6 months after surgery. To assess the nutritional status of the patients, we collect blood laboratory data, bioimpedance analysis for each visit.
  Interventions: Behavioral: Digital lifestyle management
- Non-digital lifestyle management group (No Intervention): In the control group (Non-digital lifestyle management group), 26 patients are randomly assigned to the control group (Non-digital lifestyle management group). The patients follow conventional postoperative care protocol after total thyroidectomy for thyroid cancer without using Noom application. All patients are given questionnaires to evaluate the quality of life at the baseline, 4 months, and 6 months after surgery. To assess the nutritional status of the patients, we collect blood laboratory data, bioimpedance analysis for each visit.

INTERVENTIONS:
Behavioral: Digital lifestyle management — Digital lifestyle management for Weight Loss Control after Thyroidectomy
  Arms: Digital lifestyle management group

SUMMARY:
Thyroid hormones play an important role in the regulation of the body's metabolism. But the relationship between thyroid hormone status and the basal metabolism rate is not absolute. Because thyroid hormone function is not the only factor of control the metabolism and it can be influenced by various factors such as physical activity and diet.

Weight change after thyroidectomy is one of the concerns for thyroid cancer patients. The evidence on the bodyweight changes following thyroidectomy has not been established well. Being overweight and obese can increase the risk of developing many potential health problems, such as heart disease, diabetes, high blood pressure, and malignant disease.

Recently, digital health care technology has been developed and applied for medical purposes in many clinical practices. Digital Lifestyle Management is one of the strategies that can be helpful for the obese to control their body weight by lifestyle modification. It provides comprehensive, multifactorial, intensive interventions which are delivered via the digital health care mobile service Noom application.

The aim of this study is to evaluate the efficacy of digital lifestyle management on body weight and quality of life after total thyroidectomy in thyroid cancer patients by using the digital health care Noom application.

DETAILED DESCRIPTION:
The present study is a prospective randomized control trial. A total of 80 patients who underwent total thyroidectomy for thyroid cancer is included. Fifty-four patients are randomly assigned to the digital lifestyle management group and the other 26 patients are assigned to the non-digital lifestyle management group.

In the experimental group (digital lifestyle management group), the patients will use this application for the first 4 months with Noom applications with 1:1 personalized coaching intervention, and then, use this app by self-help program without coaching intervention. The digital lifestyle management program will record the patient's meals, exercise, steps taken, reading articles, and give feedback to each patient. In order to monitor the psychological state and quality of life of the patients, online questionnaires will be provided.

In the control group (non-digital lifestyle management group), the patients will get the conventional postoperative care protocol without using the Noom application. To investigate the weight change and quality of life, variables are collected at baseline, 4 months, and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Target: Among the patients who have undergone thyroidectomy, patients who are interested in weight management and can use the Noom app by themselves or with the help of neighbors.
* The patient has 23 or more BMI at the time of enrollment.
* In The Situational Motivation Scale (SIMS), a total of five stages of synchronization level of 68 or higher, which is the top 40% of the 112 points (1st stage: pre-consumption stage; stage 2: deliberation stage; stage 3: preparation stage; stage 4: action stage)
* The patient agreed about participating in this study.

Exclusion Criteria:

* The patient was diagnosed with chronic diseases (hepatic disease, kidney disease, diabetes, etc.).
* In the case where there is no member who can support among family members,
* The patient who is not a smartphone or has difficulty using digital technology.
* When it is difficult to lose weight (pregnancy and pregnancy preparation, breastfeeding, and less than 12 months after childbirth)
* If the patient has a history of psychiatric illness (eating disorder, depression, etc.).
* If the patient is taking diet-related drugs or health supplements, or treatments.
* If there is a restriction on physical activity (not allowed to exercise for more than 30 minutes a day).

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Weight change | baseline, 4 months, 6 months
  Change from baseline weight at 4 months and 6 months after surgery

SECONDARY OUTCOMES:
Changes of results about questionnaires for quality of life (Korean Obesity Quality of Life (KOQOL)) | baseline, 4 months, 6 months
  Change from baseline results of questionnaires at 4 months and 6 months after surgery
  # Korean Obesity Quality of Life (KOQOL)
  * Range: 4-60
  * Higher scores: impaired QOL
Changes of results about questionnaires for quality of life (World Health Organization Quality of Life - Brief Form (WHOQOL-Bref)) | baseline, 4 months, 6 months
  Change from baseline results of questionnaires at 4 months and 6 months after surgery
  # World Health Organization Quality of Life - Brief Form (WHOQOL-Bref)
  * Range: 0-100
  * Higher scores: higher QOL
Changes of results about questionnaires for quality of life (Pittsburgh Sleep Quality Index (PSQI)) | baseline, 4 months, 6 months
  Change from baseline results of questionnaires at 4 months and 6 months after surgery
  # Pittsburgh Sleep Quality Index (PSQI)
  * Range: 0-21
  * Lower scores: a healthier sleep quality
Changes of results about questionnaires for quality of life (Korean-Beck Depression Inventory-II (K-BDI-II)) | baseline, 4 months, 6 months
  Change from baseline results of questionnaires at 4 months and 6 months after surgery
  # Korean-Beck Depression Inventory-II (K-BDI-II)
  * Range: 0-63
  * Higher scores: Depression
Changes of results about questionnaires for quality of life (State-Trait Anxiety Inventory (STAI)) | baseline, 4 months, 6 months
  Change from baseline results of questionnaires at 4 months and 6 months after surgery
  # State-Trait Anxiety Inventory (STAI)
  * Range: 20-80
  * Higher scores: anxiety
Changes of results about questionnaires for quality of life (Rosenberg Self-Esteem Scale (RSES)) | baseline, 4 months, 6 months
  Change from baseline results of questionnaires at 4 months and 6 months after surgery
  # Rosenberg Self-Esteem Scale (RSES)
  * Range: 0-30
  * Higher scores: lower self-esteem
Changes of results about questionnaires for quality of life (Body Shape Questionnaire (BSQ-8C) ) | baseline, 4 months, 6 months
  Change from baseline results of questionnaires at 4 months and 6 months after surgery
  # Body Shape Questionnaire (BSQ-8C)
  * Range: 8-48
  * Higher values: body dissatisfaction
Changes of results about questionnaires for quality of life (Dutch Eating Behaviour Questionnaire (DEBQ)) | baseline, 4 months, 6 months
  Change from baseline results of questionnaires at 4 months and 6 months after surgery
  # Dutch Eating Behaviour Questionnaire (DEBQ)
  * Range: 33-165
  * Higher scores: the eating behavior
Changes of waist circumstance | baseline, 4 months, 6 months
  Waist circumstance difference
Changes of hip circumstance | baseline, 4 months, 6 months
  Hip circumstance difference
Changes of body fat percent | baseline, 4 months, 6 months
  Body fat percent difference
Changes of lean body mass | baseline, 4 months, 6 months
  Lean body mass difference
Changes of total cholesterol level | baseline, 4 months, 6 months
  Biological index
Changes of HDL cholesterol level | baseline, 4 months, 6 months
  Biological index
Changes of LDL cholesterol level | baseline, 4 months, 6 months
  Biological index
Changes of triglyceride level | baseline, 4 months, 6 months
  Biological index
Changes of aspartate aminotransferase (AST) level | baseline, 4 months, 6 months
  Biological index
Changes of alanine aminotransferase (ALT) level | baseline, 4 months, 6 months
  Biological index
Changes of gamma-glutamyl transferase (GGT) level | baseline, 4 months, 6 months
  Biological index
Changes of free T3 level | baseline, 4 months, 6 months
  Biological index
Changes of free T4 level | baseline, 4 months, 6 months
  Biological index
Changes of TSH level | baseline, 4 months, 6 months
  Biological index

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Eun Lee, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea